CLINICAL TRIAL: NCT03142399
Title: Effect of Supplementation With Whey Protein in Preservation of Muscle Mass and Strength, Quality of Life of Patients With Heart Failure in Cardiac Rehabilitation
Brief Title: Effect of Whey Protein' Supplementation and Exercise in Patients With Heart Failure
Acronym: PROT-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Elisa Maia dos Santos, Master on Cardiovascular Sciences, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Whey Protein NICBrazil
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure; Sarcopenia; Muscle Loss; Quality of Life
Keywords: heart failure; cardiac reabilitation; nutritional status; quality of life; milk protein
MeSH Terms: conditions — Heart Failure; Sarcopenia; Muscular Atrophy | interventions — Whey Proteins; Dietary Supplements; Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whey protein (Experimental): The whey protein group will receive whey protein supplementation 30g/day of whey protein during three months (12 weeks)
  Interventions: Dietary Supplement: whey protein
- placebo group (Placebo Comparator): The placebo group (maltodextrin) will receive 30g/day of maltodextrin during three months (12 weeks)
  Interventions: Dietary Supplement: whey protein

INTERVENTIONS:
Dietary Supplement: whey protein — Supplementation with whey protein isolate or maltodextrin (30 grams per day) for 12 weeks associated with supervised exercise and nutritional counseling in patients with heart failure.
  Other Names: supplementation with milk protein

SUMMARY:
The aim of this study is evaluate the effect of whey protein supplementation on muscle mass preservation, improvement of strength and quality of life, and inflammatory parameters in patients with heart failure NYHA I or II followed by a cardiac rehabilitation program.

DETAILED DESCRIPTION:
Heart failure is the final route of most heart diseases and is a worldwide problem due to its high prevalence, morbidity and mortality. In Brazil, it is an important cause of hospitalization and one of the most important health challenges, since its prevalence tends to increase with the aging of the population and the increase in the survival of patients who have suffered acute coronary events. This is an ongoing epidemic problem, resulting in a high socioeconomic cost, represented by the expense of medications, repeated hospitalizations, loss of productivity, early retirements, possible surgeries and, ultimately, heart transplantation. In this sense, it is of great importance to carry out studies that evaluate the possible benefits of new clinical and nutritional interventions for HF patients, favoring the development of treatment strategies for these individuals and also for public health.

Our hypothesis is based on the fact that whey protein supplementation associated with physical exercise in patients with heart failure could promote preservation of muscle mass, increase in muscle strength, and improve quality of life, Body composition and physical capacity. The volunteers will receive 30 grams per day of whey protein or maltodextrin in a double-blind, controlled clinical trial lasting 12 weeks. During this period they will perform supervised physical exercise 3 times a week in a cardiac rehabilitation program. They will also receive nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure NYHA I or II after medical evaluation;
* Indication to participate in a cardiac rehabilitation program;
* Fully medicated for heart disease;
* Age greater than or equal to 50 years;
* Ejection fraction less than 50%.

Exclusion Criteria:

* Neoplasia at any site;
* Impaired renal function (<50ml / min / 1.73m2);
* Impaired hepatic function (TGP> 150U / l) or decompensated hepatic cirrhosis classified with Child-Pugh B or C;
* Presence of ressincronizer or other device;
* Atrial fibrilation;
* Allergy of milk protein.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Preservation of skeletal muscle mass | 12 weeks
  Assessment of body composition through bioelectrical impedance and anthropometry

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  Evaluation of health-related quality of life through the application of the Minnesota Living With Heart Failure Questionnaire validated for brazilian population
Muscle strength | 12 weeks
  Evaluation of manual gripping force through dynamometry
Change in peak oxygen uptake (VO2 peak) | 12 weeks
  Cardiopulmonary exercise test will be performed to measure VO2 peak and other parameters representative of cardiovascular reserve.
Microvascular reactivity | 12 weeks
  A laser speckle contrast imaging system with a laser wavelength of 785 nm (PeriCam PSI system, Perimed, Järfälla, Sweden) coupled to iontophoresis of acetylcholine and sodium nitroprusside will measure non-invasively real time cutaneous microvascular flow changes in the forearm. For the post occlusive reactive hyperemia (PORH) test, arterial occlusion will be performed with suprasystolic pressure (50 mmHg above the systolic arterial pressure) using a sphygmomanometer applied to the arm of the subject over three minutes. Peak skin flow will be measured after pressure release.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lorenzo, PhD, Study Director — National Institute of Cardiology, Laranjeiras, Brazil; Annie SB Moreira, PhD, Study Director — National Institute of Cardiology, Laranjeiras, Brazil
Locations (1):
- Elisa Maia dos Santos, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
All volunteer information obtained during the collection, intervention and data analysis will not be available other researchers.

REFERENCES:
- [Derived] Dos Santos EM, de Moraes R, Tibirica EV, Huguenin GVB, Moreira ASB, De Lorenzo AR. Whey protein supplementation for the preservation of mass and muscular strength of patients with heart failure: study protocol for a randomized controlled trial. Trials. 2018 Aug 8;19(1):431. doi: 10.1186/s13063-018-2811-4. PMID 30089525